CLINICAL TRIAL: NCT00622492
Title: ECMO in Newborn Infants: Circulatory Changes in Relation to Venovenous and Venoarterial Bypass. Implications for Peripheral Organ Circulation
Brief Title: Circulatory Changes During Venovenous (VV)- and Venoarterial (VA) Extracorporeal Membrane Oxygenation (ECMO)
Acronym: ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: V. Christmann, Radboud University Nijmegen Medical Centre
Other Study IDs: 2007/219
Record Dates: First submitted 2008-01-30; First posted 2008-02-25 (Estimated); Last update posted 2008-02-25 (Estimated); Status verified 2008-02

CONDITIONS: Pulmonary Hypertension of the Newborn (PPHN)
Keywords: VV-ECMO; VA-ECMO; PPHN; organ circulation
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, urine

GROUPS / COHORTS (2):
- VV-ECMO: newborn infants with reversible causes of PPHN eligible for ECMO treatment
  Interventions: Other: echocardiography Doppler sonography, blood and urine sampling
- VA-ECMO: newborn infants with reversible causes of PPHN eligible for ECMO treatment
  Interventions: Other: echocardiography Doppler sonography, blood and urine sampling

INTERVENTIONS:
Other: echocardiography Doppler sonography, blood and urine sampling — data registration and collection at standard intervals from directly before cannulation until 24 hours after decannulation from ECMO

SUMMARY:
Rationale: Persistent pulmonary hypertension of the newborn (PPHN) is a life threatening disease with a high mortality rate. Extracorporeal Membrane Oxygenation (ECMO) with veno-arterial (V-A) or veno-venous (V-V) cannulation can provide a last treatment option. Differences in circulatory changes between V-A and V-V ECMO concerning the course of PPHN and organ perfusion are not known. Independent of the underlying disease, courses of ECMO runs (with both systems) may differ a lot. Impairment of pulmonary and renal function and oedema is frequently seen. Mechanisms that may play a role are not well understood yet. A better understanding of hemodynamic changes in systemic and pulmonary circulation during treatment of PPHN with ECMO as well as consecutive changes in organ perfusion and function will help to develop more rationalistic treatment strategies to accelerate the recovery to a normal neonatal circulation and shorten ECMO treatment. This will reveal positive effects for patients as well as favourable effects on economic aspects for this very intensive treatment.

Primary objective: I.Evaluation of changes in pulmonary and systemic circulation during VV- ECMO treatment and difference between V-V- and V-A ECMO Secondary objectives:II.Evaluation of changes in cerebral, renal and mesenterial organ perfusion during ECMO treatment and difference between V-V- and V-A ECMO III.Evaluation of hemodynamic changes during ECMO treatment in relation to renal function and difference between V-V- and V-A ECMO IV.Evaluation of BNP as diagnostic parameter regarding fluid homeostasis during ECMO treatment and difference between V-V- and V-A ECMO Study design: observational; including two cohorts. The first cohort consists of a group of patients that have been evaluated in a former study, exclusively treated with V-A ECMO. The second cohort of patients will prospectively include patients receiving V-V as well as V-A ECMO. A study period:2 and a half years. All consecutively admitted patients for ECMO treatment at the department of neonatology of the RUNMC will be evaluated for inclusion into the study. Study population: Inclusion: Newborn infants with gestational age older than 34 weeks and reversible causes of PPHN eligible for ECMO treatment. Exclusion:Newborn infants with congenital diaphragmatic hernia, other congenital malformations and post-cardiosurgery.

Intervention: Standard treatment following the ECMO protocol of the department; evaluation at standard intervals starting directly before cannulation for ECMO until 24 hours after decannulation:registration of hemodynamic variables,parameters for organ perfusion using echocardiography and Doppler sonography, blood and urine sampling and registration of physiological and patient data.

Main study parameters/endpoints: Assessment of:Hemodynamic changes in pulmonary and systemic circulation Secondary and other parameters/endpoints:

Assessment of:Changes in cerebral, renal and mesenterial blood flow, renal function in relation hemodynamic changes,BNP in relation to fluid homeostasis

ELIGIBILITY:
Inclusion Criteria:

* Reversible cause of PPHN
* Newborn infant
* Older 34 weeks gestational age

Exclusion Criteria:

* Congenital diaphragmatic hernia
* Congenital malformation
* Post-cardiosurgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: newborn infants with PPHN admitted to the NICU Radboud University Medical Centre for ECMO treatment consecutive patient sampling
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Background] Tanke RB, Daniels O, van Lier HJ, van Heyst AF, Festen C. Neonatal pulmonary hypertension during extracorporeal membrane oxygenation. Cardiol Young. 2000 Mar;10(2):130-9. doi: 10.1017/s1047951100006594. PMID 10817297